CLINICAL TRIAL: NCT06516926
Title: An Open-label, Randomized, Multi-center Phase II Clinical Study of SHR-4602 for Injection in Subjects With HER2-expressing or -Mutated Unresectable or Metastatic Solid Tumors
Brief Title: SHR-4602 for Injection in Subjects With HER2-expressing or -Mutated Unresectable or Metastatic Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4602-201
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: HER2-expressing or -Mutated Unresectable or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Experimental)
  Interventions: Drug: SHR-4602
- Dose 2 (Experimental)
  Interventions: Drug: SHR-4602
- Dose 3 (Experimental)
  Interventions: Drug: SHR-4602

INTERVENTIONS:
Drug: SHR-4602 — Intravenous infusion, cycle every 21 days;

SUMMARY:
This is an open-label, randomized, multi-center phase II study to evaluate the safety, tolerability, PK, and efficacy of SHR-4602 monotherapy in subjects with HER2-expressing or -mutated unresectable or metastatic solid tumors.

During the study, a safety monitoring committee (SMC), consisting of the principal investigator, sponsor representative, etc., will be established to review data from the study regarding safety, PK, efficacy, etc. The SMC will make decisions on study-related issues.

The study includes a screening period (begins when the informed consent form (ICF) is signed and ends at the first dose), a treatment period (from the first dose to the last dose), and a follow-up period (end-of-treatment safety follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years (inclusive);
2. ECOG PS of 0 or 1;
3. Subjects are willing to provide tumor tissue samples for immunohistochemistry, ISH, or genetic testing to confirm HER2 expression or mutation; the sponsor on the enrollment;
4. Have at least one measurable lesion according to RECIST v1.1;
5. Expected survival ≥ 3 months;
6. Major organ functions meet the following criteria ；
7. Female subjects of childbearing potential must agree to take contraceptive measures, and use acceptable contraceptive measures with their partners from the signing of the ICF to 8 months after the last dose (see 13.1.2 for details); female subjects must have a negative serum pregnancy test within 7 days prior to the first dose, be non-lactating, and agree to avoid egg donation during the treatment period until 8 months after the last dose of the investigational drug;
8. Male subjects with female partners of childbearing potential must agree to use acceptable contraceptive measures during the treatment period until 8 months after the last dose of the investigational drug (see 13.1.2 for details), and agree not to donate sperm during this period. Male subjects whose partner has become pregnant must use condoms, and no other contraceptive methods are required;
9. Voluntarily participate in this clinical study, be willing and able to comply with procedures related to clinical visits and study, and understand and have signed the informed consent.

Exclusion Criteria:

1. Active brain metastases, carcinomatous meningitis, or primary central nervous system (CNS) tumors that have not been treated with surgery or radiotherapy; s
2. subjects with peripheral neuropathy (those with mild symptoms that do not require treatment and not affect the study results or increase the risk may be included as judged by the investigator);
3. Have received surgery (major surgery for cancer), chemotherapy, molecular targeted therapy, immunotherapy, cell therapy, or radiotherapy within 4 weeks prior to the first dose (palliative radiotherapy within 2 weeks prior to the first dose);
4. Are participating in another clinical study or have received the last dose in a clinical study less than 4 weeks from the first dose;
5. Have received treatment with strong CYP3A inducers or inhibitors, or P-gp inhibitors or inducers within 5 half-lives prior to the first dose;
6. Subjects with toxicities and/or complications from prior treatment that have not recovered to NCI-CTCAE Grade ≤ 1 may be enrolled if the investigator judges that these conditions are of NCI-CTCAE Grade ≤ 2 and no safety risk to the subjects;
7. Have the following lung diseases or medical history: (1) known or suspected interstitial lung disease; (2) moderate to severe lung diseases that seriously affect lung function within the past 3 months, including but not limited to idiopathic pulmonary fibrosis, organizing pneumonia/obliterative bronchiolitis, pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease (COPD), and obstructive/restrictive lung disease, which may interfere with the testing or management of treatment-related pulmonary toxicities; (3) any autoimmune, connective tissue, or inflammatory disease involving the lungs, such as rheumatoid arthritis, Sjögren's syndrome, and sarcoidosis; (4) prior pneumonectomy; (5) Grade ≥ 3 interstitial lung disease during prior treatment with immune checkpoint inhibitors. Subjects with interstitial lung changes may be enrolled if there is no safety risk as judged by the investigator;
8. Have had pleural fluid, ascites, or pericardial effusion requiring intervention within 2 weeks prior to the first dose;
9. Have active autoimmune disease, disease requiring treatment with systemic steroids or immunosuppressive drugs, other acquired (HIV infection) or congenital immunodeficiency, or history of organ transplantation (including allogeneic bone marrow transplantation);
10. Have poorly controlled or severe cardiovascular and cerebrovascular diseases, including but not limited to: (1) acute coronary syndrome, congestive heart failure (New York Heart Association [NYHA] Cardiac Function Class ≥ II), or aortic dissection within 6 months prior to the first dose of the investigational product; (2) new-onset severe/unstable angina within the past 2 months; (3) myocardial ischemia requiring long-term medication and NYHA Class ≥ II cardiac insufficiency; (4) acute myocardial infarction within 6 months before screening; (5) supraventricular arrhythmia or ventricular arrhythmia requiring treatment or interventions; (6) cerebrovascular accidents (transient ischemic attack, cerebral hemorrhage, or stroke) and pulmonary embolism within 6 months prior to the first dose of the investigational drug;
11. Known hereditary or acquired hemorrhage and thrombophilia (such as hemophilia and coagulopathy);
12. Have untreated active hepatitis (active hepatitis B, defined as hepatitis B virus surface antigen [HBsAg] positive and HBV-DNA ≥ 500 IU/mL; active hepatitis C, defined as hepatitis C virus antibody [HCV-Ab] positive and HCV-RNA above the lower limit of detection);
13. Have experienced severe infection within 30 days prior to the first dose, including but not limited to infection complications, bacteremia, and severe pneumonia requiring hospitalization; have experienced active infection treated with therapeutic intravenous antibiotics within 2 weeks prior to the first dose. subjects who have received prophylactic antibiotic therapy (e.g., for prevention of urinary tract infection) can be enrolled;
14. Other malignancies within the past 5 years or currently, except for cured cervical carcinoma in situ and basal or squamous cell carcinoma of skin;
15. Known to be allergic to any component or excipient of the SHR-4602 product, or have a history of severe anaphylaxis to other monoclonal antibody/fusion protein drugs; Have other severe physical or psychiatric disorders or laboratory abnormalities, which may increase the risk of participating in this study or interfere with the study results, as well as other conditions that make subjects unsuitable for participating in this study as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Two years objective response rate (ORR); | Two years

SECONDARY OUTCOMES:
Duration of response (dor) | Two years
Progression-free survival (PFS) | Two years
Best overall response (BOR) | Two years
Disease control rate (DCR) | Two years
Incidence and severity of adverse events (aes) | Two years
Severe adverse events (saes) (graded as per CTCAE v5.0) | Two years
Blood concentrations of conjugated antibodies | Two years
Blood concentrations of total antibodies | Two years
Blood concentrations of free toxin. | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided